CLINICAL TRIAL: NCT01749514
Title: A Phase 2, Open Label, Ascending Dose Study of ACE-536 for the Treatment of Anemia in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS)
Brief Title: Study of Luspatercept for the Treatment of Anemia in Patients With Myelodysplastic Syndrome (MDS) (MK-6143-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A536-03; MK-6143-001 (Other: Merck); A536-03 (Other: Acceleron); 2012-002523-14 (EudraCT Number)
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Anemia
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Luspatercept 0.125mg/kg (Cohort 1) (Experimental): Participants receive luspatercept 0.125mg/kg as a subcutaneous (SC) injection every 3 weeks (Q3W) on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 0.25mg/kg (Cohort 2) (Experimental): Participants receive luspatercept titrated up to 0.25mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 0.50mg/kg (Cohort 3) (Experimental): Participants receive luspatercept titrated up to 0.50mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 0.75mg/kg (Cohort 4) (Experimental): Participants receive luspatercept titrated up to 0.75mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 1.00mg/kg (Cohort 5) (Experimental): Participants receive luspatercept titrated up to 1.00mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 1.33mg/kg (Cohort 6) (Experimental): Participants receive luspatercept titrated up to 1.33mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Luspatercept 1.75mg/kg (Cohort 7) (Experimental): Participants receive luspatercept titrated up to 1.75mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: Luspatercept
- Expansion Cohort (Experimental): Participants receive an initial dose of luspatercept 1.0mg/kg SC on Day 1 of the Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated via Fibonacci scheme up to a maximum dose of 1.75mg/kg based on the safety review team (SRT) recommendations
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Participants receive luspatercept up to 1.75mg/kg subcutaneously (SC) every 3 weeks for up to 5 cycles (each cycle length = 21 days).
  Other Names: MK-6143; A536

SUMMARY:
The purpose of this study is to evaluate the effects of luspatercept (MK-6143, formerly called ACE-536) on anemia in patients with low or intermediate-1 risk myelodysplastic syndrome (MDS). There is no primary hypothesis in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of idiopathic/de novo myelodysplastic syndrome (MDS) or non-proliferative chronic myelomonocytic leukemia (CMML), according to WHO criteria (white blood count, 13,000/uL), that meets International Prognostic Scoring System (IPSS) classification of low or intermediate-1 risk disease as determined by microscopic and standard cytogenetic analyses of the bone marrow and peripheral complete blood count (CBC) obtained during screening
* Anemia defined as:

  * Mean hemoglobin concentration <10.0 g/dL of 2 measurements (one performed within one day prior to Cycle 1 Day 1 and the other performed 7-28 days prior to Cycle 1 Day 1, not influenced by red blood cell (RBC) transfusion within 7 days of measurement for non-transfusion dependent patients (defined as having received <4 units of RBCs within 8 weeks prior to Cycle 1 Day 1), or Transfusion dependent, defined as having received ≥4 units of RBCs within 8 weeks prior to Cycle 1 Day 1
* Serum erythropoietin levels and prior erythropoiesis-stimulating agent (ESA) treatment:
* Dose escalation cohorts and expansion cohort 1 patients: Serum erythropoietin level >500 U/L, OR, if ≤500 U/L, patient is non-responsive, refractory, or intolerant to erythropoiesis-stimulating agents (ESAs), or ESAs are contraindicated or unavailable
* Expansion cohort 2 patients: If patient is RS+ (defined as having ≥15% ring sideroblasts in the bone marrow), no prior ESA treatment and serum erythropoietin level ≤ 200 U/L. If a patient is RS- (defined as having <15% ring sideroblasts in the bone marrow), prior ESA treatment and any serum erythropoietin level is allowed
* No alternative treatment options, per applicable MDS guidelines, are available and/or appropriate for the patient, at the discretion of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (if related to anemia).
* Adequate renal (creatinine ≤2 x upper limit of normal [ULN]) and hepatic (total bilirubin <2 x ULN and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 x ULN) function
* Adequate transferrin saturation (≥15%), ferritin (≥ 50 µg/L), folate (≥4.5 nmol/L [≥2.0 µg/L]) and vitamin B12 (≥148 pmol/L [≥ 200 pg/mL]) during screening (supplementation and retest during screening is acceptable)
* Females of child bearing potential (defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy, or are not naturally postmenopausal ≥24 consecutive months) must have negative urine or blood pregnancy test prior to enrollment and use adequate birth control methods (abstinence, oral contraceptives, barrier method with spermicide, or surgical sterilization) during study participation and for 12 weeks following the last dose of luspatercept. Males must agree to use a latex condom during any sexual contact with females of child-bearing potential while participating in the study and for 12 weeks following the last dose of luspatercept, even if he has undergone a successful vasectomy. Patients must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of luspatercept
* Patients are able to adhere to the study visit schedule, understand and comply with all protocol requirements
* Patients understand and are able to provide written informed consent

Key Exclusion Criteria:

* Prior treatment with azacitidine or decitabine
* Treatment within 28 days prior to Cycle 1 Day 1 with:

  * Erythropoiesis stimulating agent (ESA)
  * Granulocyte colony-stimulating factor (G-CSF) and granulocyte-macrophage colony stimulating factor (GM-CSF)
  * Lenalidomide
* Iron chelation therapy if initiated within 56 days prior to Cycle 1 Day 1
* Treatment with another investigational drug or device, or approved therapy for investigational use ≤28 days prior to Cycle 1 Day 1, or if the half-life of the previous product is known, within 5 times the half-life prior to Cycle 1 Day 1, whichever is longer
* Major surgery within 28 days prior to Cycle 1 Day 1. Patients must have completely recovered from any previous surgery prior to Cycle 1 Day 1
* Platelet count <30 x 109/L.
* Any active infection requiring parenteral antibiotic therapy within 28 days prior to Cycle 1 Day 1 or oral antibiotics within 14 days of Cycle 1 Day 1
* History of stroke, deep venous thrombosis (DVT) or arterial embolism within 6 months prior to Cycle 1 Day 1
* Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B (HBV) or active infectious hepatitis C (HCV)
* Any malignancy other than MDS which has not been in remission and/or has required systemic therapy including radiation, chemotherapy, hormonal therapy or surgery, within the last year prior to Cycle 1 Day 1
* Uncontrolled hypertension, defined as systolic blood pressure (BP) ≥ 150 mm Hg or diastolic BP ≥ 100 mm Hg
* Pregnant or lactating females
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational drug
* Any other condition not specifically noted above which, in the judgment of the investigator, would preclude the patient from participating in the study
* Transfusion event within 7 days prior to Cycle 1 Day 1
* Prior treatment with sotatercept (MK-7962, formerly called ACE-011) or luspatercept.
* Secondary MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Acceleron Investigative Site, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Platzbecker U, Gotze KS, Kiewe P, Germing U, Mayer K, Radsak M, Wolff T, Chromik J, Sockel K, Oelschlagel U, Haase D, Illmer T, Al-Ali HK, Silling G, Reynolds JG, Zhang X, Attie KM, Shetty JK, Giagounidis A. Long-Term Efficacy and Safety of Luspatercept for Anemia Treatment in Patients With Lower-Risk Myelodysplastic Syndromes: The Phase II PACE-MDS Study. J Clin Oncol. 2022 Nov 20;40(33):3800-3807. doi: 10.1200/JCO.21.02476. Epub 2022 Aug 23. PMID 35998303
- [Derived] Platzbecker U, Germing U, Gotze KS, Kiewe P, Mayer K, Chromik J, Radsak M, Wolff T, Zhang X, Laadem A, Sherman ML, Attie KM, Giagounidis A. Luspatercept for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes (PACE-MDS): a multicentre, open-label phase 2 dose-finding study with long-term extension study. Lancet Oncol. 2017 Oct;18(10):1338-1347. doi: 10.1016/S1470-2045(17)30615-0. Epub 2017 Sep 1. PMID 28870615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 116 participants were enrolled and received treatment.
Groups:
- Luspatercept 0.125mg/kg (Cohort 1): Participants received luspatercept 0.125mg/kg as a subcutaneous (SC) injection every 3 weeks (Q3W) on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.25mg/kg (Cohort 2): Participants received luspatercept titrated up to 0.25mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.50mg/kg (Cohort 3): Participants received luspatercept titrated up to 0.50mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.75mg/kg (Cohort 4): Participants received luspatercept titrated up to 0.75mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.00mg/kg (Cohort 5): Participants received luspatercept titrated up to 1.00mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.33mg/kg (Cohort 6): Participants received luspatercept titrated up to 1.33mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.75mg/kg (Cohort 7): Participants received luspatercept titrated up to 1.75mg/kg via Fibonacci scheme, SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Expansion Cohort: Participants received an initial dose of luspatercept 1.0mg/kg SC on Day 1 of the Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated via Fibonacci scheme up to a maximum dose of 1.75mg/kg based on the safety review team (SRT) recommendations.
Period: Overall Study
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Started | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
Completed | 3 | 3 | 3 | 6 | 3 | 5 | 3 | 82
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (19.1) | 59.0 (27.8) | 66.3 (5.1) | 64.8 (11.3) | 73.7 (3.8) | 68.2 (7.1) | 63.7 (19.6) | 71.6 (9.6) | 70.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 0 | 1 | 2 | 30 | 44
  Male | 0 | 0 | 1 | 3 | 3 | 5 | 1 | 59 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 3 | 6 | 3 | 5 | 3 | 80 | 105
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 9 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89 | 116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion Status [Count of Participants; unit: Participants] — Low Transfusion Burden (LTB) participants are defined as those who received <4 units of red blood cells (RBCs) within 8 weeks prior to baseline (Cycle 1 Day 1). High Transfusion Burden (HTB) participants are defined as those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline.
  Participants
    HTB | 2 | 2 | 3 | 3 | 3 | 6 | 1 | 31 | 51
    LTB | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 58 | 65
Hemoglobin level [Mean (Standard Deviation); unit: g/dl] — Hemoglobin level of participants in peripheral blood was reported. Population: All enrolled participants with baseline hemoglobin level data available. Data were not collected from 3 participants at baseline.
  g/dl
    number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 5 | 3 | 87 | 113
    (all) | 10.30 (0.98) | 8.91 (0.81) | 8.83 (0.31) | 8.55 (0.75) | 8.37 (1.10) | 8.42 (0.58) | 9.53 (0.06) | 8.79 (1.01) | 8.81 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Low Transfusion Burden (LTB) Participants With Modified Erythroid Response (mHI-E)
Description: The mHI-E for LTB participants was defined as a hemoglobin increase of ≥1.5 g/dL from baseline for ≥14 days or rolling 2 weeks (in the absence of red blood cell [RBC] transfusions). Hemoglobin measurements within 7 days following RBC transfusion were excluded from analysis. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. Rolling 2 weeks was defined as any consecutive 2 weeks during the study. The percentage of LTB participants with mHI-E were reported.
Time Frame: Any consecutive 2 weeks during the study (up to approximately 75 weeks)
Population: All enrolled LTB participants who received at least one dose of luspatercept and received <4 units of RBCs within 8 weeks prior to baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 58
Percentage of participants | 0 [0 to 97.5] | 0 [0 to 97.5] |  | 66.7 [9.4 to 99.2] |  |  | 100 [15.8 to 100] | 69.0 [55.5 to 80.5]

2. Primary Outcome: Percentage of High Transfusion Burden (HTB) Participants With mHI-E
Description: The mHI-E for HTB participants was defined as a ≥4 units or ≥50% reduction in RBC transfusion burden during any rolling 8-week window compared to baseline. HTB participants were those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline. Rolling 8 weeks was defined as any consecutive 8 weeks during the study. The percentage of HTB participants with mHI-E were reported.
Time Frame: Any consecutive 8 weeks during the study (up to approximately 75 weeks)
Population: All enrolled HTB participants who received at least one dose of luspatercept and who required ≥4 units of RBC transfusions within 8 weeks prior to baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 6 | 1 | 31
Percentage of Participants | 50.0 [1.26 to 98.7] | 50.0 [1.26 to 98.7] | 33.3 [0.84 to 90.6] | 33.3 [0.84 to 90.6] | 33.3 [0.84 to 90.6] | 50.0 [11.8 to 88.2] | 100 [2.5 to 100] | 54.8 [36.0 to 72.7]

3. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 24 weeks
Population: All enrolled participants who received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
Participants | 1 | 2 | 3 | 5 | 3 | 4 | 2 | 75

4. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To an AE
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 12 weeks
Population: All enrolled participants who received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

5. Secondary Outcome: Rate of Erythroid Response (HI-E) Per International Working Group (IWG) 2006 Response Criteria
Description: Per IWG 2006 response criteria, rate of HI-E is defined as the percentage of participants for whom the mean of all hemoglobin value from baseline during any rolling 8-week increased ≥1.5 g/dL in the absence of transfusion for LTB participants, or a reduction by ≥4 units of RBCs transfusion over any rolling 8-week window for HTB patients. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. HTB participants were those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline. Rolling 8 weeks was defined as any consecutive 8 weeks during the study.
Time Frame: Any consecutive 8 Weeks during the study treatment (up to approximately 75 weeks)
Population: All enrolled participants who received at least one dose of luspatercept.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
Percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 33.3 [4.3 to 77.7] | 33.3 [0.8 to 90.6] | 50.0 [11.8 to 88.2] | 100 [29.2 to 100] | 53.9 [43.0 to 64.6]

6. Secondary Outcome: Rate of Platelet Response (HI-P) Per IWG 2006 Criteria
Description: Per IWG 2006 response criteria, HI-P was defined for participants with baseline value ≥20 x 10^9/L as the platelet increase in any rolling 8 weeks ≥30 x 10^9 and for participants with baseline value <20 x 10^9/L as the platelet increase in any rolling 8 weeks >20 x 10^9/L with increase of at least 100%. The rolling 8-week was defined as any consecutive 8 weeks during the study. The percentage of participants with HI-P were reported.
Time Frame: Any consecutive 8 Weeks during the study treatment (up to approximately 75 weeks)
Population: All enrolled participants who received at least one dose of luspatercept and had baseline platelet count <100x10^9/L.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 17
Percentage of participants |  |  | 0 (0.0) [0.0 to 97.5] |  | 0 (0.0) [0.0 to 84.2] | 0 (0.0) [0.0 to 97.5] |  | 23.5 (6.8) [6.8 to 49.9]

7. Secondary Outcome: Rate of Neutrophil Response (HI-N) Per IWG 2006 Criteria
Description: Per IWG 2006 response criteria, HI-N was defined as the neutrophil increase in any rolling 8 weeks is at last 100% and an absolute increase > 0.5 x 10^9/L. The rolling 8-week was defined as any consecutive 8 weeks during the study. The percentage of participants with HI-N response were reported.
Time Frame: Any consecutive 8 Weeks during the study treatment (up to approximately 75 weeks)
Population: All enrolled participants who received at least one dose of luspatercept and had baseline neutrophil count <1.0×10^9/L.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 18
Percentage of Participants | 0 [0.0 to 97.5] |  | 100 [2.5 to 100] | 0 [0.0 to 97.5] |  | 66.7 [9.4 to 99.2] | 100 [2.5 to 100] | 25.0 [8.7 to 49.1]

8. Secondary Outcome: Duration of HI-E Per IWG 2006 Response Criteria
Description: Per IWG 2006 response criteria, duration of HI-E response was defined as the time from the first day of the first rolling 8-week interval of showing response to the last day of the last consecutive rolling 8-week interval of showing response. HI-E response for LTB participants was defined as hemoglobin increase ≥ 1.5 g/dL during any rolling 8-week window and for HTB HI-E was defined as RBC transfusion reduction ≥4 units during any rolling 8 weeks. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. HTB participants were those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline. The rolling 8-week was defined as any consecutive 8 weeks during the study.
Time Frame: up to approximately 75 weeks
Population: All enrolled participants who received at least one dose of luspatercept. Per protocol, the participants with response were pooled into low and high dose groups to increase the accuracy of the analyses.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Low Dose Luspatercept 0.125-0.5 mg/kg (Cohorts 1, 2, 3): Participants received luspatercept 0.125mg/kg up to 0.5mg/kg as a SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days)
- High Dose Luspatercept 0.75-1.75mg/kg (Cohorts 4, 5, 6, 7 & Expansion): Participants receive luspatercept 0.75mg/kg up to 1.75mg/kg as a SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
Arm/Group | Low Dose Luspatercept 0.125-0.5 mg/kg (Cohorts 1, 2, 3) | High Dose Luspatercept 0.75-1.75mg/kg (Cohorts 4, 5, 6, 7 & Expansion)
Number analyzed (Participants) | 9 | 107
Days | 78 (7.8) | 88 (22.8)

9. Secondary Outcome: Time to HI-E Per IWG 2006 Response Criteria
Description: Per IWG 2006 response criteria, the time to HI-E response was defined as the first date of the rolling 8-week interval of showing response minus first dose date plus 1. HI-E response for LTB participants was defined as hemoglobin increase ≥ 1.5 g/dL during any rolling 8 weeks window and for HTB HI-E was defined as RBC transfusion reduction ≥4 units during any rolling 8 weeks. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. HTB participants were those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline. The rolling 8-week was defined as any consecutive 8 weeks during the study.
Time Frame: Any consecutive 8 weeks during the study (up to approximately 75 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low Dose Luspatercept 0.125-0.5 mg/kg (Cohorts 1, 2, 3) | High Dose Luspatercept 0.75-1.75mg/kg (Cohorts 4, 5, 6, 7 & Expansion)
Number analyzed (Participants) | 9 | 107
Days | 35 (48.1) | 17 (18.3)

10. Secondary Outcome: Mean Change From Baseline to Day 113 in Frequency of RBC Transfusions
Description: Frequency of RBC transfusion was defined as the total number of RBC transfusions received. Per protocol, the mean change from baseline to Day 113 in frequency of RBC transfusion was reported in the HTB participants (those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline).
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of RBC transfusions
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 6 | 1 | 31
Number of RBC transfusions
  Baseline | 2.50 (0.71) | 2.50 (2.12) | 4.00 (0.00) | 2.00 (0.00) | 4.00 (1.00) | 2.83 (0.75) | 3.00 (NA) — NA = SD could not be calculated due to low number of participants with RBC transfusion. | 3.06 (1.34)
  Baseline to Day 113 | -0.70 (0.71) | 0.11 (0.69) | 0.38 (2.08) | 0.40 (2.12) | -0.31 (1.21) | -0.36 (1.03) | -2.46 (NA) — NA = SD could not be calculated due to low number of participants with RBC transfusion. | -0.85 (1.14)

11. Secondary Outcome: Rate of RBC Transfusion Independence (RBC-TI)
Description: Rate of RBC-TI was defined as percentage of participants with ≥2 units of RBC transfusions at baseline who experienced transfusion independence which was defined as ≥8 weeks without a transfusion while on treatment. Per protocol, rate of RBC-TI was reported in HTB participants (those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline).
Time Frame: Up to approximately 16 weeks
Population: All enrolled HTB participants who received at least one dose of luspatercept and had ≥2 units of RBC transfusions at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 3 | 6 | 1 | 57
Percentage of participants | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 66.7 [22.3 to 95.7] | 0 [0.0 to 70.8] | 33.3 [4.3 to 77.7] | 100 [2.5 to 100] | 43.9 [30.7 to 57.6]

12. Secondary Outcome: Time to Maximum Concentration (Tmax) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of Tmax. Tmax was defined as time to the maximum concentration of luspatercept reached. Tmax was based on non-compartmental analysis and a mean Tmax value was presented.
Time Frame: Cycle 1 Day 1: Predose, Cycle 1: Days 8, 11, 15: Postdose; Cycle 2 Day 1, Cycle 2 Day 8, Cycle 4 Day 1, Cycle 5 Day 1, and Cycle 5 Days 8, 15: Postdose (each cycle length = 21 days)
Population: All participants who have received at least one dose of luspatercept and had sufficient pharmacokinetic samples collected and assayed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
Days | 9.93 (35.73) | 7.23 (20.68) | 10.16 (39.56) | 7.16 (5.46) | 7.23 (20.68) | 8.47 (31.58) | 6.65 (8.92) | 7.77 (21.76)

13. Secondary Outcome: Terminal Half-Life (t ½) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of t½. t½ was defined as the time required to divide the luspatercept plasma concentration by two after reaching pseudo-equilibrium, following a single dose of luspatercept. t½ was based on non-compartmental analysis and a mean t1/2 value was presented.
Time Frame: as for outcome 12
Population: All participants who received at least one dose of luspatercept and had sufficient pharmacokinetic samples collected and assayed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 5 | 1 | 62
Days | 23.78 (22.29) | 9.15 (44.83) | 15.14 (5.94) | 14.45 (16.02) | 13.75 (7.37) | 14.76 (24.43) | 26.56 (9.19) | 14.74 (44.35)

14. Secondary Outcome: Maximum Concentration (Cmax) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of Cmax. Cmax was defined as the maximum concentration of luspatercept reached. Cmax was based on non-compartmental analysis and a mean Cmax value was presented.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 89
ug/mL | 0.64 (34.88) | 0.96 (92.99) | 2.33 (27.16) | 3.76 (42.29) | 4.35 (12.87) | 7.46 (14.55) | 9.66 (7.52) | 5.73 (26.93)

15. Secondary Outcome: Area Under the Concentration-Time Curve of Luspatercept From Time 0 to Day 21 (AUC0-21)
Description: Blood samples were collected at specified intervals for the determination of AUC0-21. AUC0-21 was defined as the area under the concentration-time curve of luspatercept from time zero to Study Day 21. AUC0-21 was based on non-compartmental analysis and a mean AUC0-21 value was presented.
Time Frame: Cycle 1 Day 1: Predose, Cycle 1 Days 8, 11, 15 and Cycle 2 Day 1: Postdose (each cycle length = 21 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/m
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 2 | 6 | 3 | 6 | 3 | 87
day*ug/m | 9.29 (32.16) | 12.56 (94.99) | 36.90 (4.19) | 51.82 (35.93) | 62.46 (25.20) | 112.56 (17.00) | 137.56 (1.13) | 80.02 (27.77)

16. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Iron
Description: Blood samples were to be collected at pre-specified time intervals to determine serum iron concentration. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: No data were collected for the percent change from baseline to day 113 in concentration of serum iron.
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percent Change From Baseline to Day 113 in Total Iron Binding Capacity (TIBC)
Description: Blood samples were collected at pre-specified time intervals to determine TIBC. The percentage change from baseline in TIBC was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for TIBC.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 5 | 2 | 86
Percent change | -1.49 (8.940) | 1.61 (1.392) | -6.70 (6.050) | 10.91 (11.806) | 7.46 (11.727) | -12.27 (22.144) | -4.16 (2.435) | -2.40 (9.916)

18. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Transferrin
Description: Blood samples were to be collected at pre-specified time intervals to determine concentration of transferrin. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: No data were collected for the percent change from baseline to day 113 in concentration of transferrin.
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Soluble Transferrin Receptor
Description: Blood samples were collected at pre-specified time intervals to determine soluble transferrin receptor concentration. The percentage change from baseline in concentration of soluble transferrin receptor was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for soluble transferrin receptor.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 2 | 2 | 5 | 0 | 5 | 2 | 77
Percent change | 60.88 (76.427) | -31.46 (5.135) | -4.62 (6.527) | 36.35 (21.718) |  | -17.11 (32.861) | 19.25 (7.793) | 35.35 (44.228)

20. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Ferritin
Description: Blood samples were collected at pre-specified time intervals to determine serum ferritin concentration. The percentage change from baseline in concentration of serum ferritin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for serum ferritin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 5 | 2 | 87
Percent change | -19.55 (32.845) | 58.63 (24.342) | 74.31 (160.308) | 1.16 (23.487) | 19.38 (25.666) | 8.56 (41.532) | -16.07 (27.172) | -1.51 (46.269)

21. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Non-Transferrin Bound Iron (NTBI)
Description: Blood samples were to be collected at pre-specified time intervals to determine concentration of NTBI. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: No data were collected for the percent change from baseline to day 113 in concentration of NTBI.
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Hepcidin
Description: Blood samples were collected at pre-specified time intervals to determine soluble hepcidin concentration. The percentage change from baseline in concentration of soluble hepcidin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for serum hepcidin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 5 | 1 | 64
Percent change | -42.40 (5.907) | 6.56 (35.740) | -14.55 (39.855) | -15.62 (20.814) | -5.54 (49.144) | 65.41 (179.249) | -64.51 (NA) — NA = SD could not be calculated due to low number of participants with hepcidin values | 30.15 (143.118)

23. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Erythropoietin
Description: Blood samples were collected at pre-specified time intervals to determine serum erythropoietin concentration. The percentage change from baseline in concentration of serum erythropoietin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All participants who received at least one dose of luspatercept and had data available for serum erythropoietin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 5 | 2 | 84
Percent change | 144.48 (232.336) | 110.51 (85.751) | 122.85 (163.500) | 1.81 (48.208) | 749.10 (902.000) | 146.49 (160.087) | 29.07 (80.426) | 238.85 (974.226)

24. Secondary Outcome: Percent Change From Baseline to Day 113 in Reticulocyte Count
Description: Blood samples were collected at pre-specified time intervals to determine reticulocyte count. The percentage change from baseline in mean reticulocyte count was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for reticulocyte count.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 1 | 2 | 5 | 3 | 3 | 2 | 74
Percent change | 110.82 (127.489) | 8.10 (NA) — NA=SD could not be calculated due to insufficient number of participants in the study. | 79.77 (45.816) | 28.29 (28.434) | 76.16 (54.003) | 0.45 (19.770) | 84.06 (108.298) | 41.37 (73.445)

25. Secondary Outcome: Percent Change From Baseline to Day 113 in Direct Bilirubin Level
Description: Blood samples were collected at pre-specified time intervals to determine serum direct bilirubin concentration. The percentage change from baseline in mean concentration direct bilirubin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for direct bilirubin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 3 | 1 | 64
Percent change | -18.45 (6.569) | 12.38 (38.465) | 2.33 (NA) — NA = SD could not be calculated due to low number of participants with direct bilirubin values | 7.22 (20.592) | -5.00 (NA) — NA = SD could not be calculated due to low number of participants with direct bilirubin values | -7.41 (12.830) | 6.78 (NA) — NA = SD could not be calculated due to low number of participants with direct bilirubin values | -0.50 (27.541)

26. Secondary Outcome: Percent Change From Baseline to Day 113 in Total Bilirubin Level
Description: Blood samples were collected at pre-specified time intervals to determine total bilirubin concentration. The percentage change from baseline in mean concentration total bilirubin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for total bilirubin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 5 | 2 | 85
Percent change | -25.41 (5.596) | 4.32 (26.094) | 47.43 (51.076) | 4.02 (10.439) | -25.08 (17.240) | -25.84 (19.893) | 10.68 (20.258) | 13.26 (37.239)

27. Secondary Outcome: Percent Change From Baseline to Day 113 in Lactate Dehydrogenase Level
Description: Blood samples were collected at pre-specified time intervals to determine serum lactate dehydrogenase level. The percentage change from baseline in mean concentration lactate dehydrogenase level was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for lactate dehydrogenase.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 5 | 2 | 85
Percent change | 13.09 (28.850) | -10.28 (6.589) | 0.03 (32.694) | 2.76 (7.848) | -15.20 (25.355) | -2.52 (18.669) | -11.91 (35.318) | 20.58 (46.589)

28. Secondary Outcome: Percent Change From Baseline to Day 113 in Nucleated RBC (nRBC)
Description: Blood samples were to be collected at pre-specified time intervals to determine concentration of nRBC. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: No data were collected for the percent change from baseline to day 113 in concentration of nRBC.
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Bone-Specific Alkaline Phosphatase (BSAP)
Description: Blood samples were collected at pre-specified time intervals to determine serum BSAP concentration. The percentage change from baseline in concentration BSAP was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for BSAP.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 3 | 5 | 1 | 23
Percent change | -6.41 (3.698) | -36.70 (9.430) | -24.60 (16.413) | 47.48 (42.431) | 14.15 (13.191) | -6.43 (25.559) | 15.27 (NA) — NA = SD could not be calculated due to low number of participants with BSAP values | 8.31 (23.800)

30. Secondary Outcome: Percent Change From Baseline to Day 113 in Concentration of Serum Cross-Linked C-Telopeptide of Type I Collagen (CTX)
Description: Blood samples were collected at pre-specified time intervals to determine serum CTX. The percentage change from baseline in concentration of CTX was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 113
Population: All enrolled participants who received at least one dose of luspatercept and had data available for CTX.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.125mg/kg (Cohort 1) | Luspatercept 0.25mg/kg (Cohort 2) | Luspatercept 0.50mg/kg (Cohort 3) | Luspatercept 0.75mg/kg (Cohort 4) | Luspatercept 1.00mg/kg (Cohort 5) | Luspatercept 1.33mg/kg (Cohort 6) | Luspatercept 1.75mg/kg (Cohort 7) | Expansion Cohort
Number analyzed (Participants) | 1 | 0 | 1 | 5 | 3 | 4 | 1 | 24
Percent change | -4.42 (NA) — NA = SD could not be calculated due to low number of participants with CTX values |  | 16.26 (NA) — NA = SD could not be calculated due to low number of participants with CTX values | 26.37 (24.669) | 15.94 (35.018) | 13.04 (62.513) | -70.97 (NA) — NA = SD could not be calculated due to low number of participants with CTX values | 22.66 (51.177)

ADVERSE EVENTS:
Time Frame: Up to approximately 75 weeks
Description: All-cause mortality was reported on all enrolled participants. Serious and non-serious AEs were reported among participants who received at least one dose of study treatment.
Groups:
- Luspatercept 0.125 mg/kg (Cohort 1): Participants received luspatercept 0.125mg/kg as a subcutaneous (SC) injection every 3 weeks (Q3W) on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days)
- Luspatercept 0.25 mg/kg (Cohort 2): Participants received luspatercept titrated up to 0.25mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.50 mg/kg (Cohort 3): Participants received luspatercept titrated up to 0.50mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.75 mg/kg (Cohort 4): Participants received luspatercept titrated up to 0.75mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.0 mg/kg (Cohort 5): Participants received luspatercept titrated up to 1mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.33 mg/kg (Cohort 6): Participants received luspatercept titrated up to 1.33mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.75 mg/kg (Cohort 7): Participants received luspatercept titrated up to 1.75mg/kg SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Expansion Cohort: Participants received an initial dose of luspatercept 1mg/kg SC on Day 1 of the Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated up to a maximum dose of 1.75mg/kg based on the safety review team (SRT) recommendations.
Arm/Group | Luspatercept 0.125 mg/kg (Cohort 1) | Luspatercept 0.25 mg/kg (Cohort 2) | Luspatercept 0.50 mg/kg (Cohort 3) | Luspatercept 0.75 mg/kg (Cohort 4) | Luspatercept 1.0 mg/kg (Cohort 5) | Luspatercept 1.33 mg/kg (Cohort 6) | Luspatercept 1.75 mg/kg (Cohort 7) | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/6 | 0/3 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/6 | 1/3 | 3/6 | 1/3 | 14/89
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/3 | 5/6 | 3/3 | 3/6 | 2/3 | 62/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.125 mg/kg (Cohort 1) (N=3) | Luspatercept 0.25 mg/kg (Cohort 2) (N=3) | Luspatercept 0.50 mg/kg (Cohort 3) (N=3) | Luspatercept 0.75 mg/kg (Cohort 4) (N=6) | Luspatercept 1.0 mg/kg (Cohort 5) (N=3) | Luspatercept 1.33 mg/kg (Cohort 6) (N=6) | Luspatercept 1.75 mg/kg (Cohort 7) (N=3) | Expansion Cohort (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.125 mg/kg (Cohort 1) (N=3) | Luspatercept 0.25 mg/kg (Cohort 2) (N=3) | Luspatercept 0.50 mg/kg (Cohort 3) (N=3) | Luspatercept 0.75 mg/kg (Cohort 4) (N=6) | Luspatercept 1.0 mg/kg (Cohort 5) (N=3) | Luspatercept 1.33 mg/kg (Cohort 6) (N=6) | Luspatercept 1.75 mg/kg (Cohort 7) (N=3) | Expansion Cohort (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 11 (12)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 11 (12)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 5 (9)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (7)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 9 (12)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 19 (25)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication or disclosure of study results will be permitted as per the agreement between the sponsor and the investigator(s).

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT01749514/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT01749514/SAP_001.pdf